CLINICAL TRIAL: NCT02704377
Title: Quality of Life and Supportive Care Preferences Following Radiation Therapy in Prostate Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Brian Focht, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-15049; NCI-2015-01289 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2015-08-31; First posted 2016-03-10 (Estimated); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Prostate Carcinoma
Keywords: Prostate Cancer Survivor
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Absorptiometry, Photon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (1):
- Supportive care (quality of life, supportive care preferences) (Experimental): Participants complete questionnaires about quality of life and preferences for supportive care treatment, wear accelerometerundergo heart rate variability(HRV) testing over 10-15 minutes while both lying down and standing, complete a walking test, wear an accelerometer for a period of 1 week, and undergo a single Dual X-ray Absorptiometry (iDXA) scan over 10 minutes. Other interventions include: Laboratory Biomarker Analysis, Quality-of-Life Assessments, and othe Questionnaire Administration.
  Interventions: Other: Undergo HRV and wear accelerometer to assess therapy complications; Procedure: Dual X-ray Absorptiometry; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Undergo HRV and wear accelerometer to assess therapy complications — Wear accelerometer undergo heart rate variability(HRV) testing over 10-15 minutes while both lying down and standing, complete a walking test, wear an accelerometer for a period of 1 week
Procedure: Dual X-ray Absorptiometry — Undergo iDXA
  Other Names: BMD scan; bone mineral density scan; DEXA; DEXA scan; dual energy x-ray absorptiometric scan; Dual Energy X-ray Absorptiometry; Dual X-Ray Absorptometry; DXA; DXA SCAN
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This pilot clinical trial studies quality of life and supportive care preferences following radiation therapy in prostate cancer survivors. Studying quality of life and supportive care preferences in patients undergoing radiation therapy may help identify the effects of treatment on patients with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To develop an understanding of the impacts of prostate cancer on aspects of psychological stress, physiological stress and health related quality of life (HRQL) for men who are being treated with some level of radiation therapy (RT).

II. To gain insight into the perceived needs of survivors depending on their disease stage, treatment regimen and side effects.

SECONDARY OBJECTIVES:

I. To explore whether biomarkers of stress, inflammation and autonomic control (heart rate variability [HRV]) can confirm or dispel the self-reported measures of psychological distress and HRQL of a unique population of aging men with prostate cancer.

OUTLINE:

Participants complete questionnaires about quality of life and preferences for supportive care treatment, undergo heart rate variability testing over 10-15 minutes while both lying down and standing, complete a walking test, wear an accelerometer for a period of 1 week, and undergo a single intelligent dual-energy X-ray absorptiometry (iDXA) scan over 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Diagnosis of prostate cancer
* Treatment with primary radiation (brachytherapy or external beam therapy), radiation + androgen deprivation therapy (ADT) or salvage prostatectomy
* Body mass index (BMI) (26 - 40 kg/m^2)
* Treating oncologist consent
* Ambulatory or able to engage in walking for at least 45 minutes per intervention visit
* Sedentary lifestyle, as engaging in less than 100 minutes structured aerobic walking, cycling or swimming per week

Exclusion Criteria:

* Poor diagnosis or other cancer
* Severe heart or systemic disease: evidence of documented myocardial infarction, chronic unstable angina, symptomatic congestive heart failure, uncontrolled hypertension
* Severe musculoskeletal disease: severe muscle or joint disorders due to disease or trauma, amputations, or any condition that significantly impair physical capabilities, as defined by the physician
* Non-ambulatory
* Concurrent diagnosis of organic brain syndrome, dementia, mental retardation, or significant sensory deficit
* Major mental illness (e.g., schizophrenia, major depressive disorder)
* Unwilling to give consent

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-05-08 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Develop an understanding of the impacts of prostate cancer on HRQL measured by the SF-36 | Baseline
  Significance tests for the difference between treatment groups on all primary outcomes will be conducted. Data will be individually standardized by covariates such as age, disease stage and grade, time on treatment values and will be evaluated using an analysis of co-variance statistical mode. Descriptive statistics for the feasibility measures will be calculated prospectively throughout the trial.
Psychological resiliency measured by Connor Davidson Resiliency Scale | Baseline
  The relationship with self-reported measures of quality of life and stress will be determined. Significance tests for the difference between treatment groups on all primary outcomes will be conducted. Data will be individually standardized by covariates such as age, disease stage and grade, time on treatment values and will be evaluated using an analysis of co-variance statistical mode. Descriptive statistics for the feasibility measures will be calculated prospectively throughout the trial.
Explore whether heart rate variability is associated with the SF-36 and Connor Davidson Resiliency Scale. | Up to 1 week
  Significance tests for the difference between treatment groups on all primary outcomes will be conducted. Data will be individually standardized by covariates such as age, disease stage and grade, time on treatment values and will be evaluated using an analysis of co-variance statistical mode. Descriptive statistics for the feasibility measures will be calculated prospectively throughout the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Focht, PhD, FACSM, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu